CLINICAL TRIAL: NCT04440462
Title: Lingual Frenulotomy in the Newborn: a Randomized Clinical Trial to Evaluate the Analgesic Effect of a Water and Sugar Solution in a Minor Surgical Procedure
Brief Title: Analgesia in Lingual Frenulotomy in the Newborn
Acronym: RE-GLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 13/2019
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Frenulum Breve
Keywords: Ankyloglossia; Frenulotomy; water and sugar solution
MeSH Terms: conditions — Ankyloglossia | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugar and water solution (Experimental): 2 ml of a water and sugar solution (3 full-teaspoons of granulated sugar dissolved in half glass of water)
  Interventions: Other: Sugar and water solution
- Sterile water (Active Comparator): 2 ml of sterile water
  Interventions: Other: Sterile water

INTERVENTIONS:
Other: Sugar and water solution — 2 ml of a water and sugar solution (3 full-teaspoons of granulated sugar dissolved in half glass of water)
  Arms: Sugar and water solution
Other: Sterile water — 2 ml of sterile water
  Arms: Sterile water

SUMMARY:
Ankyloglossia (tongue-tie) is a congenital anomaly characterized by a short lingual frenulum that limits the physiological tongue movement and occurs with an estimated prevalence between 4 and 10% of the newborns. This condition can be associated with difficulty in breastfeeding which can be painful for the mother, dysfunctional swallowing and future speech difficulties. The prevalence of nipple pain among women breastfeeding newborns with ankyloglossia is estimated to be between 36 and 80%. Since an early intervention can prevent the difficulties that may occur during the child's growth and can also improve the mothers and patients' quality of life, it is important to evaluate the lingual frenulum in the first days of life. The treatment of ankyloglossia consists in the frenulotomy which allows the release of the lingual frenulum and is a relatively simple procedure with few side effects and minimal post-operative. Different methods performed with or without local anaesthesia by means of scissors, blade, laser (etc.) are described in literature for the procedure the newborn.

The hypothesis of the study is that the addition of a water and sugar solution to the standard analgesia with lidocaine may lead to a greater benefit in terms of pain control and determine the activation of different brain areas.

The primary aim of the study is to evaluate whether the administration of a water and sugar solution to newborns undergoing frenulotomy receiving topical lidocaine as standard analgesic protocol, may lead to an additional benefit in terms of pain reduction evaluated according to the Neonatal Infant Pain Scale (NIPS).

The secondary aim of the study is to evaluate through a Hitachi multichannel near-infrared spectroscopy (NIRS) the effects of the addition of a water and sugar solution to the standard analgesic protocol with topical lidocaine on the cortical activation.

ELIGIBILITY:
Inclusion Criteria

1. Term newborns (37 - 41 weeks of gestational age) within the first 10 days of life;
2. Birth weight ≥ 2500 grams;
3. Presence of ankyloglossia;
4. Indication to the frenulotomy according to the Hazelbaker Assessment Tool for Lingual Frenulum Function (HATLFF): anatomical-functional evaluation with a score lower than 8.

Exclusion Criteria:

1. Syndromic diagnosis (genetic/hereditary);
2. Pathology of main organ (heart disease, brain disease etc.);
3. Drugs intake that may interfere with the collected data (sedatives).

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 30 seconds after the frenulotomy
  The perception of pain in newborns will be evaluated according to the Internationally Validated Neonatal Infant Pain Scale (NIPS).This scale detects the presence of six behavioral expression signs of neonatal pain (facial expression, crying, respiratory pattern, arms and legs' activity, arousal state) and ranges from 0 (absence of pain) to 7 (maximal pain level).

SECONDARY OUTCOMES:
Pain reduction | During the frenulotomy
  The perception of pain in newborns will be evaluated according to the Internationally Validated Neonatal Infant Pain Scale (NIPS).This scale detects the presence of six behavioral expression signs of neonatal pain (facial expression, crying, respiratory pattern, arms and legs' activity, arousal state) and ranges from 0 (absence of pain) to 7 (maximal pain level).
Cortical oxy-haemoglobin change | 30 seconds after the frenulotomy
  Multichannel near-infrared spectroscopy will be used to estimate cerebral cortex activation by measuring increase in cortical oxy-haemoglobin (HbO2) (Hitachi multichannel NIRS system)

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Chermetz, DDS MSc, Principal Investigator — Institute for maternal and child health Burlo Garofolo; Milena Cadenaro, DDS MSc PhD, Study Director — Institute for maternal and child health Burlo Garofolo; Chiara Navarra, DDS MSc PhD, Principal Investigator — Institute for maternal and child health Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS Burlo Garofolo-, Trieste, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No